CLINICAL TRIAL: NCT02367235
Title: Analysis of Robotic Procedural Times Using the Colpassist Vaginal Positioning Device for Robotic-Assisted Sacrocolpopexy; a Randomized Controlled Trial
Brief Title: Analysis of Procedural Times Using Colpassist for Robotic-Assisted Sacrocolpopexy; a Randomized Controlled Trial
Acronym: ACRAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Boston Scientific Corporation (Industry); Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-1834
Record Dates: First submitted 2014-12-09; First posted 2015-02-20 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Pelvic Organ Prolapse
Keywords: robotic; sacrocolpopexy; Colpassist; vaginal positioning device
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional vaginal positioning device (Experimental): Patients will undergo their robotic-assisted sacrocolpopexy using a vaginally placed endo anal sizer.
  Interventions: Procedure: Traditional vaginal positioning device
- Colpassist vaginal positioning device (Experimental): Patients will undergo their robotic-assisted sacrocolpopexy using a vaginally placed Colpassist vaginal manipulator.
  Interventions: Procedure: Colpassist vaginal positioning device

INTERVENTIONS:
Procedure: Traditional vaginal positioning device — A vaginally placed endo-anal sizer will be used to position the vagina during surgery.
  Arms: Traditional vaginal positioning device
Procedure: Colpassist vaginal positioning device — A vaginally placed Colpassist will be used to position the vagina during surgery.
  Arms: Colpassist vaginal positioning device

SUMMARY:
The purpose of this study is to evaluate the efficiency of the Colpassist vaginal positioning device during robotic-assisted sacrocolpopexy.

DETAILED DESCRIPTION:
The purpose of this research study is to evaluate the efficiency of the Colpassist (Boston Scientific, Natick, MA) vaginal positioning device used during robotic-assisted sacrocolpopexy. Traditionally, vaginal positioning during robotic-assisted sacrocolpopexy is done using a device that was not designed specifically for sacrocolpopexy, commonly a vaginally placed endo anal sizer. It is possible the Colpassist device will result in shorter operative times because Colpassist is flat which makes it easier to sew against. Also, the width of the device is designed to be similar to the width of the vagina which should improve visibility during surgery.

Enrolled patients will be randomized to undergo their planned robotic-assisted sacrocolpopexy using either a vaginally placed endo anal sizer or a vaginally placed Colpassist vaginal positioning device. Both surgeon and patient will be blinded to which device was used at the time of surgery. Length of time to complete each step of the sacral colpoexy that involves use of a vaginal positioning device (dissection of the anterior and posterior vaginal walls, attachment of anterior and posterior vaginal mesh, attachment of sacral mesh) will be recorded during the surgery to measure operative efficiency. Surgeon and surgical-assistant satisfaction will be recorded with each device.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old
* Planned robotic-assisted sacrocolpopexy
* English speaking
* Prior hysterectomy (either total or supra-cervical)

Exclusion Criteria:

* Age less than 18 years old
* Non-English speaking
* Pregnant women, or women desiring future pregnancy
* Planned concomitant hysterectomy

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-01; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Comparison of duration of surgical steps during sacral colpopexy | Intraoperative
  Length of time will be recorded for each step of the sacral colpopexy that utilizes the vaginal positioning device (dissection of anterior vaginal wall, dissection of posterior vaginal wall, attachment of anterior vaginal mesh, attachment of posterior vaginal mesh, and attachment of sacral mesh) during the surgery. No follow up will be required by the patient.

SECONDARY OUTCOMES:
Surgeon and surgical-assistant satisfaction with the device | On the day of surgery
  Surgeon and surgical assistant satisfaction will be assessed via questionnaire immediately after surgery. No follow up will be required of the surgeons or the assistants.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Geller, MD, Principal Investigator — UNC-Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill - Female Pelvic Medicine and Reconstructive Surgery, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No